CLINICAL TRIAL: NCT02900807
Title: CT-scan Airways Mensuration - Correlation to External Measurements
Acronym: AIRWAY
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GTR_2014_24
Record Dates: First submitted 2016-09-07; First posted 2016-09-14 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-02

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Oro-tracheal intubation is performed daily in anesthesia and in the ICU. When a patient is intubated, the endotracheal tube must be inserted into the trachea to the right depth. If the tube is not deep Inserted enough there is a risk of accidental extubation and trauma to the vocal cords by the balloon. If the tube is inserted too far there is a risk of selective intubation into the right or left mainstem bronchus, which can lead to contralateral lung atelectasis and hypoxemia.

The purpose of this study is to determine whether there is a correlation between the measurement of the airway of an adult population and criteria that would be easily accessible in daily clinical practice: the height of the patient and the size of their feet.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for a CT-scan including the airways and the upper part of the chest at least until the carina
* patient size between between 150 cm and 195 cm

Exclusion Criteria:

* significant deformity of the cervical spine to accurately measure the size of patients (kyphoscoliosis...)
* impossibility of reliably know the size of the patient
* history of pharyngo-laryngeal surgery resulting in a significant deformity or a loss of anatomical landmarks incompatible with reliable measurements between dental arches and glottic plan (total laryngectomy...)
* history of lung surgery not allowing reliable location of the carina (pneumonectomy, double-lung transplant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for a CT-scan including the airways and the upper part of the chest until the hull
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
size of the patients and/or size of their feet | Duration of the CT-scan : about 1 hour
  measured with a height chart and/or a pedometer
measurement of patients' airways | Duration of the CT-scan : about 1 hour
  Mensurations of airways measured on imaging (CT-scan)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Taylor, MD, Study Director — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France